CLINICAL TRIAL: NCT05486182
Title: Impact of 18F-fluoroestradiol (FES) Positron Emission Tomography (PET) on the Therapeutic Treatment of Metastatic Breast Cancer Patients, Initially ER Positive and HER2 Negative, in Relapse After First-line Therapy Combining Hormone Therapy
Brief Title: Impact of 18F-FES PET on the Therapeutic Treatment of Patients With Metastatic Breast Cancer
Acronym: ESTROTIMP
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: Simbec-Orion Group (Industry); Keosys (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ZX-2021-FES-ESTROTIMP-4; 2021-003601-21 (EudraCT Number); 2024-517400-11-00 (EU CTIS Number)
Record Dates: First submitted 2022-03-04; First posted 2022-08-03 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prospective population (Experimental)
  Interventions: Drug: 18F Fluoroestradiol Radiopharmaceutical with PET/CT

INTERVENTIONS:
Drug: 18F Fluoroestradiol Radiopharmaceutical with PET/CT — Administration of one dose of 18F FES for PET/CT imaging
  Other Names: ESTROTEP

SUMMARY:
This is a multi-center study in France to evaluate the impact of ESTROTEP PET/CT results on the therapeutic management of patients with metastatic breast cancer (MBC).

Each patient will be screened to determine whether the patient meets all the inclusion criteria and none of the exclusion criteria.

After inclusion, a standardized pre ESTROTEP PET/CT questionnaire will be completed by the investigators to evaluate the initial management plan. Patient will perform the ESTROTEP PET/CT examination at visit 2. A standardized post ESTROTEP PET/CT questionnaire will then be completed by the investigators.

Patients will be followed for 12 months to evaluate their clinical status and standard of care investigations.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged at least 18 years old at the time of enrolment
2. Oestrogen-receptor positive primary breast cancer in IHC (ER ≥10%)
3. HER2-negative primary breast cancer (0, 1+, 2+ FISH negative)
4. Metastatic stage with at least one lesion identifiable on the conventional work-up other than a liver lesion
5. Patient relapsing under first-line treatment combining a CDK4/6inhibitor and hormone therapy
6. Patient having undergone an FDG PET/CT during follow-up of first-line treatment for metastatic tumour revealing the relapse or undergoing a baseline FDG PET/CT seeking the relapse during 2nd line staging (according to the recommendations of the Guide to Correct Use (GBU) for medical imaging tests). A period of 2 to 28 days will be respected between the 2 PET/CT scans (FDG/FES).
7. ECOG 0, 1 or 2
8. Life expectancy of at least 12 months
9. Patient registered with a Social Security scheme
10. Patient having signed an informed consent form
11. Patient able to follow the study procedures and fill in the quality of life questionnaires

Exclusion Criteria:

1. Isolated hepatic metastases (taking into account the high physiological hepatic uptake of FES)
2. Patients as first-line treatment for metastatic cancer or aftersecond-line treatment for metastatic cancer
3. Person presenting a known allergy to one of the components of EstroTep
4. Patients having been treated with a CDK4/6 inhibitor in combination with an SERM or SERD as first-line metastatic therapy
5. atients suffering from severe or known chronic liver or renal failure
6. Patient following a low-sodium diet or having alcohol consumption levels incompatible with the administration of EstroTep, according to the investigator's opinion
7. Woman of childbearing age with no effective means of contraception according to the investigator's opinion
8. Severe intercurrent disease or comorbidity assessed at risk
9. Persons referred to in articles L. 1121-5 to L. 1121-8 and L11222 of the French Public Health Code

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of ESTROTEP PET/CT on metastatic breast cancer patients management, initially ER+ and HER2-, in relapse after first-line treatment combining hormone therapy. | Change from baseline therapeutic measure at 15 days after ESTROTEP PET/CT
  The percentage of patients for whom a substantial therapeutic measure was implemented following an analysis of the FES PET examination. This assessment will be performed prospectively by means of a standardised questionnaire completed by the prescribing clinician, when the request for an FES PET/CT is made. The therapeutic modality initially planned and the modality actually used may be determined by a multidisciplinary consultation meeting depending on the centre. This questionnaire will completed again within a maximum period of 15 days following the FES PET/CT in order to specify the final therapeutic measure.
  Substantial measures will be considered to be any major modifications made in terms of: therapeutic modalities, diagnostic modalities and follow-up modalities.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Cochet, Principal Investigator — Centre Georges Francois Leclerc
Locations (11):
- France (11):
  - CGFL, Dijon
  - CHU Grenoble Alpes, La Tronche
  - CHU de Limoges - Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Institut du Cancer de Montpellier, Montpellier
  - Hôpital Américain de Paris, Neuilly-sur-Seine
  - Centre Antoine Lacassagne, Nice
  - Hôpital Tenon, Paris
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud
  - Institut Claudius Regaud Centre de Lutte Contre le Cancer, Toulouse